CLINICAL TRIAL: NCT06020274
Title: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, Resource (iCF-PWR) Program: How Does it Work?
Brief Title: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, Resource Program: How Does it Work?
Acronym: iCF-PWR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Authority - Regina Area (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-166
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis in Children; Siblings; Mental Health; Internet-based Intervention
Keywords: cystic fibrosis; child; adolescent; siblings; mental health; Internet-based intervention; anxiety; depression
MeSH Terms: conditions — Psychological Well-Being; Cystic Fibrosis; Anxiety Disorders; Depression | interventions — Health; Health Resources

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the iCF-PWR group or the standard care group. The investigators will follow CONSORT guidelines for non-pharmacological trials with 1:1 random assignment to iCF-PWR or standard care. As such, 30 children with CF/30 child siblings will be randomly assigned to the iCF-PWR group and 30 children with CF/30 child siblings will be randomly assigned to the standard care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iCF-PWR Program (Experimental): Parents are encouraged to review the program along with their child and then children are encouraged to complete the program 1-2 additional times (or as many times as they like). It is suggested that modules be completed at a rate of 1-2 per week, with program completion ranging from 3-6 weeks. Additional mental health resources are provided at the end of the program.
  Interventions: Behavioral: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program
- Standard Care (No Intervention): Participants will continue to receive their usual standard care related to CF (i.e., accessing services through their local health authority and CF clinic). Following the proposed maximum program completion time-frame (i.e., 6 weeks) and follow-up time period (i.e., 3 months), those in the standard care groups will be provided access to iCF-PWR.

INTERVENTIONS:
Behavioral: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program — The iCF-PWR program is a self-guided mental health prevention program designed for families with CF. Upon logging on to the iCF-PWR, the viewer will see two paths (i.e., child with CF or sibling) and will be encouraged by program narrator to choose the appropriate path. Each pathway (i.e., child with CF or sibling) is comprised of five text/voice-delivered, animated, interactive modules: (1) CF education, (2) CF health, (3) emotions and CF, (4) cognitive behaviour model of emotions, and (5) coping strategies. Each module takes 15-20 minutes to complete.
  Arms: iCF-PWR Program

SUMMARY:
The goal of the clinical trial is to test whether a mental health program that is delivered through the Internet works well for children and adolescents with cystic fibrosis (CF) and their healthy siblings. The main questions it aims to answer are:

* Does the program improve the mental health such as depression and anxiety symptoms?
* Does the program improve overall quality of life?
* Does the program improve self-efficacy - an individual's belief in their ability to complete tasks to achieve their goals?

Participants will:

* Fill out an online survey asking questions about their personal and health information, as well as their mental health before the program
* Complete the online mental health program
* Fill out an online survey asking questions about their mental health after completing the program, and 1-month and 3-months following completing the program

Participants be compared against another group of children with CF and their healthy siblings who are on a waitlist and receiving usual CF treatment. Researchers will compare participants scores before starting the program with their scores immediately following completing the program, 1-month, and 3-month after completing the program. Researchers hope to develop a program that improves mental health, quality of life, self-efficacy, and knowledge about CF.

DETAILED DESCRIPTION:
BACKGROUND: Children with cystic fibrosis (CF) and family members have been shown to experience elevated psychological symptoms, such as depression and anxiety. Over the past decade, significant advances have been made in the care of people living with CF, including major steps toward assessing and promoting emotional wellness. Despite these advances, there has been no specific mental health program designed for families with CF in Canada until recently. To address the limitations of traditionally delivered mental health programs and lack of developed Internet-delivered mental health programs for children with CF and their siblings, the investigators created the self-guided Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program for children with CF and their child siblings. The program was designed with a stepped-care model in mind, whereby all children with CF and their child siblings could access and benefit from this preventative program (i.e., least resource intensive intervention). If a child was in need of more intensive services prior to or following iCF-PWR completion, then services could be accessed through regular avenues (i.e., CF team, local outpatient/inpatient public mental health services, or private practice). The self-guided iCF-PWR program was informed by those with lived experiences with CF, the empirical literature [i.e., CF, mental health disorders in childhood and adolescence with chronic illnesses, universal mental health prevention in children and adolescence, stepped care, and team expertise. Individual contributions from specific children with CF and child siblings directed the development of individual program avatars and provided the personal stories and experiences embedded in the program modules. Preliminary evidence suggests that the program is deemed acceptable. However, to date the efficacy of the iCF-PWR is unknown.

PARTICIPANTS: G*Power 3.1 was used to calculate the study sample size based upon on our primary analyses (i.e., mixed model analysis of variance ANOVA]). Assuming 80% power, an alpha of 0.05, and effect size of 0.25 (small to medium effect), a sample size of at least 24 participants in each group would be needed. The investigators aim to recruit 30 participants per group to address attrition. 60 children (ages 8 to 12 years) with CF and 60 child siblings (ages 8 to 12 years) will be recruited from the CF clinics and CF Chapters, CF advocacy groups, advocacy groups for pediatric chronic illness across Canada in a 1-year prospective study. Participants will be randomly assigned to either the iCF-PWR group or the standard care group. The investigators will seek to have equal representation of gender across both groups. Following the proposed maximum program completion time-frame (i.e., 6 weeks) and follow-up time period (i.e., 3 months), those in the standard care groups will be provided access to iCF-PWR.

HYPOTHESES:

1. The iCF-PWR group will have significant reductions in self-reported anxiety symptoms from pre- to post-program and at follow-up time points compared to the standard care group.
2. The iCF-PWR group will have significant reductions in self-reported depressive symptoms from pre- to post-program and at follow-up time points compared to the standard care group.
3. The iCF-PWR group will have significant reductions in self-reported health anxiety from pre- to post-program and at follow-up time points compared to the standard care group.
4. The iCF-PWR group will have significant improvements in self-reported quality of life from pre- to post-program and at follow-up time points compared to the standard care group.
5. The iCF-PWR group will have significant improvements in self-reported self-efficacy from pre- to post-program and at follow-up time points compared to the standard care group.

METHODS/PROCEDURES: Parent/guardian will be provided an overview of procedure in initial email. Via Qualtrics (i.e., online survey platform) (1) parent/guardian will be asked to complete consent form/facilitate the endorsement of assent form with child and complete and complete a short personal/health demographics questionnaire about themselves and their child, and (2) their child will be asked to complete a series of self-report questionnaires assessing anxiety, depression, health anxiety, quality of life, self-efficacy, and disease knowledge (pre-program measurement). The parent caregiver will help facilitate the child's completion of questionnaires. Parent will be asked to complete measures of parent-rated child anxiety and depression. This will take 5 minutes. Via email, child and parent/guardian will be provided a link to complete these measures once the program is completed (post-program measurement) and at two follow-up time points (1 month and 3 months post-program). Measure of satisfaction will be completed by child at post-program as well. Measures will take approximately 30 to 40 minutes to complete at each time-point. Similar time-points for measure completion will be used for both study groups (i.e., iCF-PWR and standard care groups). However, the satisfaction questionnaire will not be completed by standard care group.

Parents are encouraged to review the program along with their child and then children are encouraged to complete the program at least 1 additional time, with an overall program completion ranging from 3 to 6 weeks. Children can review the program as many times as they would like. Once enrolled, parent caregiver will be provided with a username/password. Parents/participants will be instructed to keep their username/password private. They will also be encouraged to access the program in a private area, preferably in their own homes. A contact e-mail will be given for technical support and instructions on how to operate the site. All contact with the parents/participants will be via e-mail during program, although a phone number will also be provided. Inquiries via email and telephone will be fielded by study coordinator. A reminder e-mail will be sent to parents if child has not logged onto the program at least 1x/week.

ANALYSES: Statistical analyses will be performed using IBM SPSS Statistics-Version 26. Demographic data will be summarized as means and standard deviations for continuous data and frequencies for categorical data. Preliminary analyses will explore the potential impact of demographic variables (e.g., age, gender) on primary and secondary outcome variables. If demographic variables have a statistically significant impact on outcome measures, those variables will be included as covariate(s) in primary and secondary analyses. An intention-to-treat (ITT) design will be employed for all primary and secondary analyses. Primary analyses will be three 2 (group: iCF-PWR vs standard care) x 4 (time of assessment: pre-program vs. post-program vs. 1 month follow-up vs. 3 months follow-up) multi-level modeling (equivalent to mixed- model ANOVAs) to examine the effect of the intervention on the primary outcome measures (i.e., anxiety, depression, health anxiety). Secondary analyses will be two 2 (group: iCF-PWR vs standard care) x 4 (time of assessment: pre-program vs post-program vs 1 month follow-up vs 3 months follow-up) multilevel modeling to examine the effect of the intervention on the secondary outcome measures (i.e., quality of life, self-efficacy).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 8 and 12
* have a CF diagnosis or are a sibling of a child with CF
* can speak and read English. The research team does not have competence in other languages, further our program is delivered in English

Exclusion Criteria:

* have a severe cognitive impairment or a major comorbid medical or psychiatric illness, as this may impede their ability to fully participate in the program and evaluation process

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the State-Trait Anxiety Inventory for Children (STAI-C) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The STAI-C measures general anxiety in children on a continuous scale with items being rated on a 3-point Likert scale reflecting the frequency of anxiety symptom. Total scores can range from a minimum score of 20 to a maximum score of 60.
Change from Baseline in the State-Trait Anxiety Inventory for Children (STAI-C) at 1 Month | Baseline and 1-month follow up
  The STAI-C measures general anxiety in children on a continuous scale with items being rated on a 3-point Likert scale reflecting the frequency of anxiety symptom. Total scores can range from a minimum score of 20 to a maximum score of 60.
Change from Baseline in the State-Trait Anxiety Inventory for Children (STAI-C) at 3 Months | Baseline and 3-months follow up
  The STAI-C measures general anxiety in children on a continuous scale with items being rated on a 3-point Likert scale reflecting the frequency of anxiety symptom. Total scores can range from a minimum score of 20 to a maximum score of 60.
Change from Baseline in the Children's Depression Inventory-2 (CDI-2) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The CDI-2 measures cognitive, affective, and behavioural symptoms of depression in children and adolescents on a continuous scale. Each item is rated on a 3-point Likert scale ranging from 0 (absence of symptom) to 2 (definite symptom). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Children's Depression Inventory-2 (CDI-2) at 1 month | Baseline and 1-month follow up
  The CDI-2 measures cognitive, affective, and behavioural symptoms of depression in children and adolescents on a continuous scale. Each item is rated on a 3-point Likert scale ranging from 0 (absence of symptom) to 2 (definite symptom). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Children's Depression Inventory-2 (CDI-2) at 3 months | Baseline and 3-months follow up
  The CDI-2 measures cognitive, affective, and behavioural symptoms of depression in children and adolescents on a continuous scale. Each item is rated on a 3-point Likert scale ranging from 0 (absence of symptom) to 2 (definite symptom). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Childhood Illness Attitudes Scale (CIAS) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The CIAS assesses fears, beliefs, and attitudes that are associated with health anxiety and abnormal illness behaviour in school children on a continuous scale. Items are rated on a 3-point Likert scale with total scores range from 29 to 87 with higher scores reflecting higher levels of health anxiety associated behaviours.
Change from Baseline in the Childhood Illness Attitudes Scale (CIAS) at 1 month | Baseline and 1-month follow up
  The CIAS assesses fears, beliefs, and attitudes that are associated with health anxiety and abnormal illness behaviour in school children on a continuous scale. Items are rated on a 3-point Likert scale with total scores range from 29 to 87 with higher scores reflecting higher levels of health anxiety associated behaviours.
Change from Baseline in the Childhood Illness Attitudes Scale (CIAS) at 3 months | Baseline and 3-months follow up
  The CIAS assesses fears, beliefs, and attitudes that are associated with health anxiety and abnormal illness behaviour in school children on a continuous scale. Items are rated on a 3-point Likert scale with total scores range from 29 to 87 with higher scores reflecting higher levels of health anxiety associated behaviours.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL-4.0) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The PedsQL-4.0 measures health-related quality of life in healthy and acute and chronically ill children and adolescents on a continuous scale. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). The PedsQL-4.0 is comprised of four generic core scales that encompass physical functioning, emotional functioning, social functioning, and school functioning.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL-4.0) at 1 month | Baseline and 1-month follow up
  The PedsQL-4.0 measures health-related quality of life in healthy and acute and chronically ill children and adolescents on a continuous scale. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). The PedsQL-4.0 is comprised of four generic core scales that encompass physical functioning, emotional functioning, social functioning, and school functioning.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL-4.0) at 3 months | Baseline and 3-months follow up
  The PedsQL-4.0 measures health-related quality of life in healthy and acute and chronically ill children and adolescents on a continuous scale. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). The PedsQL-4.0 is comprised of four generic core scales that encompass physical functioning, emotional functioning, social functioning, and school functioning.
Change from Baseline in the Self-Efficacy Questionnaire for Children (SEQ-2) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The SEQ-C is a 21 item measures designed to assess children's perceptions of their social self-efficacy (ability to relate and get along with other peers), emotional self-efficacy (ability to regulate unpleasant emotions), and academic self-efficacy (ability to succeed in school and display appropriate learning behaviors). The three subscales each contain seven items in which participants rate their competence level on a 5-point Likert-type scale (1 = not at all to 5 = very well). Scores are summed to yield a measure of self-efficacy for each domain.
Change from Baseline in the Self-Efficacy Questionnaire for Children (SEQ-2) at 1 Month | Baseline and 1-month follow up
  The SEQ-C is a 21 item measures designed to assess children's perceptions of their social self-efficacy (ability to relate and get along with other peers), emotional self-efficacy (ability to regulate unpleasant emotions), and academic self-efficacy (ability to succeed in school and display appropriate learning behaviors). The three subscales each contain seven items in which participants rate their competence level on a 5-point Likert-type scale (1 = not at all to 5 = very well). Scores are summed to yield a measure of self-efficacy for each domain.
Change from Baseline in the Self-Efficacy Questionnaire for Children (SEQ-2) at 3 Months | Baseline and 3-months follow up
  The SEQ-C is a 21 item measures designed to assess children's perceptions of their social self-efficacy (ability to relate and get along with other peers), emotional self-efficacy (ability to regulate unpleasant emotions), and academic self-efficacy (ability to succeed in school and display appropriate learning behaviors). The three subscales each contain seven items in which participants rate their competence level on a 5-point Likert-type scale (1 = not at all to 5 = very well). Scores are summed to yield a measure of self-efficacy for each domain.
Change from Baseline in the Disease Knowledge Questionnaire at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The measure was constructed to assess CF disease knowledge as it related to the iCF-PWR content. It is comprised of 13 items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate greater CF disease knowledge.
Change from Baseline in the Disease Knowledge Questionnaire at 1 Month | Baseline and 1-month follow up
  The measure was constructed to assess CF disease knowledge as it related to the iCF-PWR content. It is comprised of 13 items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate greater CF disease knowledge.
Change from Baseline in the Disease Knowledge Questionnaire at 3 Months | Baseline and 3-months follow up
  The measure was constructed to assess CF disease knowledge as it related to the iCF-PWR content. It is comprised of 13 items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate greater CF disease knowledge.
Participants Qualitative Perception of Program Satisfaction at Week 3-6 | Week 3-6 (post-intervention)
  Six qualitative questions designed to assess participants perception of satisfaction with the iCF-PWR program. The questions directly address perceived strengths, likability, and areas of improvement for the program. Participant responses are qualitative in nature.

SECONDARY OUTCOMES:
Change from Baseline in the Children's Depression Inventory-2 - Parent Report (CDI-2 P) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The CDI-2 P assesses a parent's observation of their child's or adolescent's cognitive, affective, and behavioural symptoms of depression. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 2 (much or most of the time). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Children's Depression Inventory-2 - Parent Report (CDI-2 P) at 1 Month | Baseline and 1-month follow up
  The CDI-2 P assesses a parent's observation of their child's or adolescent's cognitive, affective, and behavioural symptoms of depression. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 2 (much or most of the time). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Children's Depression Inventory-2 - Parent Report (CDI-2 P) at 3 Months | Baseline and 3-months follow up
  The CDI-2 P assesses a parent's observation of their child's or adolescent's cognitive, affective, and behavioural symptoms of depression. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 2 (much or most of the time). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the State-Trait Anxiety Inventory - Parent Version (STAI-P) at Week 3-6 | Baseline and Week 3-6 (post-intervention)
  The STAI-P assesses state anxiety (i.e., at this present moment) in school children with and without physical symptoms. Items are rated on a 4-point Likert scale reflecting the frequency the anxiety symptom occurs (1 = not at all; 2 = sometimes; 3 = moderately; 4 = very much so). Total scores for the subscales can range from a minimum score of 20 to a maximum score of 80.
Change from Baseline in the State-Trait Anxiety Inventory - Parent Version (STAI-P) at 1 Month | Baseline and 1-month follow up
  The STAI-P assesses state anxiety (i.e., at this present moment) in school children with and without physical symptoms. Items are rated on a 4-point Likert scale reflecting the frequency the anxiety symptom occurs (1 = not at all; 2 = sometimes; 3 = moderately; 4 = very much so). Total scores for the subscales can range from a minimum score of 20 to a maximum score of 80.
Change from Baseline in the State-Trait Anxiety Inventory - Parent Version (STAI-P) at 3 Months | Baseline and 3-months follow up
  The STAI-P assesses state anxiety (i.e., at this present moment) in school children with and without physical symptoms. Items are rated on a 4-point Likert scale reflecting the frequency the anxiety symptom occurs (1 = not at all; 2 = sometimes; 3 = moderately; 4 = very much so). Total scores for the subscales can range from a minimum score of 20 to a maximum score of 80.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi D Wright, Ph.D., Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - Saskatchewan Health Authority, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quittner AL, Goldbeck L, Abbott J, Duff A, Lambrecht P, Sole A, Tibosch MM, Bergsten Brucefors A, Yuksel H, Catastini P, Blackwell L, Barker D. Prevalence of depression and anxiety in patients with cystic fibrosis and parent caregivers: results of The International Depression Epidemiological Study across nine countries. Thorax. 2014 Dec;69(12):1090-7. doi: 10.1136/thoraxjnl-2014-205983. Epub 2014 Sep 21. PMID 25246663
- [Background] Quittner AL, Abbott J, Georgiopoulos AM, Goldbeck L, Smith B, Hempstead SE, Marshall B, Sabadosa KA, Elborn S; International Committee on Mental Health; EPOS Trial Study Group. International Committee on Mental Health in Cystic Fibrosis: Cystic Fibrosis Foundation and European Cystic Fibrosis Society consensus statements for screening and treating depression and anxiety. Thorax. 2016 Jan;71(1):26-34. doi: 10.1136/thoraxjnl-2015-207488. Epub 2015 Oct 9. PMID 26452630
- [Background] Jamieson N, Fitzgerald D, Singh-Grewal D, Hanson CS, Craig JC, Tong A. Children's experiences of cystic fibrosis: a systematic review of qualitative studies. Pediatrics. 2014 Jun;133(6):e1683-97. doi: 10.1542/peds.2014-0009. PMID 24843053
- [Background] Elborn JS. Cystic fibrosis. Lancet. 2016 Nov 19;388(10059):2519-2531. doi: 10.1016/S0140-6736(16)00576-6. Epub 2016 Apr 29. PMID 27140670
- [Background] Smith BA, Georgiopoulos AM, Quittner AL. Maintaining mental health and function for the long run in cystic fibrosis. Pediatr Pulmonol. 2016 Oct;51(S44):S71-S78. doi: 10.1002/ppul.23522. PMID 27662107
- [Background] Goldbeck L, Fidika A, Herle M, Quittner AL. Psychological interventions for individuals with cystic fibrosis and their families. Cochrane Database Syst Rev. 2014 Jun 18;2014(6):CD003148. doi: 10.1002/14651858.CD003148.pub3. PMID 24941199
- [Background] Pinquart M, Shen Y. Depressive symptoms in children and adolescents with chronic physical illness: an updated meta-analysis. J Pediatr Psychol. 2011 May;36(4):375-84. doi: 10.1093/jpepsy/jsq104. Epub 2010 Nov 18. PMID 21088072
- [Background] Fauman KR, Pituch KJ, Han YY, Niedner MF, Reske J, LeVine AM. Predictors of depressive symptoms in parents of chronically ill children admitted to the pediatric intensive care unit. Am J Hosp Palliat Care. 2011 Dec;28(8):556-63. doi: 10.1177/1049909111403465. Epub 2011 Mar 30. PMID 21454321
- [Background] Moussavi S, Chatterji S, Verdes E, Tandon A, Patel V, Ustun B. Depression, chronic diseases, and decrements in health: results from the World Health Surveys. Lancet. 2007 Sep 8;370(9590):851-8. doi: 10.1016/S0140-6736(07)61415-9. PMID 17826170
- [Background] Barrett PM, Farrell LJ, Ollendick TH, Dadds M. Long-term outcomes of an Australian universal prevention trial of anxiety and depression symptoms in children and youth: an evaluation of the friends program. J Clin Child Adolesc Psychol. 2006 Sep;35(3):403-11. doi: 10.1207/s15374424jccp3503_5. PMID 16836477
- [Background] O'Donohue WT, Draper C. The case for evidence-based stepped care as part of a reformed delivery system. In Draper C, O'Donohue WT (Eds), Stepped Care and e-Health. Practical Applications to Behavioral Disorders.Springer:1-16.
- [Background] Wright KD, Switzer H, Power HA et al. Canadian research: Mental health needs of children and adolescents with CF, and their families. Presented at the Western Canadian Cystic Fibrosis Conference, Saskatoon, SK, 2020, September.
- [Background] Spielberger CD, Edwards CD, Montuori J, et al. State-Trait Anxiety Inventory for Children. Palo Alto, CA: Consulting Psychologist Press;1973.
- [Background] Kovacs M. Children's depression inventory-2. New York: Multi-Health System. 2011.
- [Background] Wright KD, Asmundson GJ. Health anxiety in children: development and psychometric properties of the Childhood Illness Attitude Scales. Cogn Behav Ther. 2003;32(4):194-202. doi: 10.1080/16506070310014691. PMID 16291551
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Muris P. A brief questionnaire for measuring self-efficacy in youths. J Psychopathol Behav Assess 2001;23:145-49.
- [Background] Shain LM, Pao M, Tipton MV, Bedoya SZ, Kang SJ, Horowitz LM, Wiener L. Comparing Parent and Child Self-report Measures of the State-Trait Anxiety Inventory in Children and Adolescents with a Chronic Health Condition. J Clin Psychol Med Settings. 2020 Mar;27(1):173-181. doi: 10.1007/s10880-019-09631-5. PMID 31127422
- [Background] Miles M, Huberman M. An Expanded Source Book: Qualitative Data Analysis. California: Sage Publications. 1994.
- [Background] Morse J, Field P. Qualitative research methods for health professionals. California: Sage Publications. 2005.